CLINICAL TRIAL: NCT04192786
Title: The Effect of Local Vibration Applied to Spastic Gastrocnemius on Muscle Architecture and Functional Properties in Multiple Sclerosis Patients
Brief Title: Local Vibration in Multiple Sclerosis Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Hacettepe University (Other)
Responsible Party: Principal Investigator, Fatma Ayvat, Research Assistant, Hacettepe University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: KA-19018
Record Dates: First submitted 2019-11-26; First posted 2019-12-10 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Multiple Sclerosis
Keywords: Multiple Sclerosis; Spasticity; Local Vibration; Muscle Architecture; Functionality
MeSH Terms: conditions — Multiple Sclerosis; Muscle Spasticity

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Treatment Group 50 Hz (Experimental)
  Interventions: Other: Standard physiotherapy program+50 Hz local vibration
- Treatment Group 100 Hz (Experimental)
  Interventions: Other: Standard physiotherapy program+100 Hz local vibration
- Control Group (Active Comparator)
  Interventions: Other: Standard physiotherapy program

INTERVENTIONS:
Other: Standard physiotherapy program+50 Hz local vibration — Standard physiotherapy program (strength, balance, gait exercises) for 50 minutes and local vibration applied to gastrocnemius (50 Hz) for 10 minutes will be performed 3 days a week for 8 weeks.
  Arms: Treatment Group 50 Hz
Other: Standard physiotherapy program+100 Hz local vibration — Standard physiotherapy program (strength, balance, gait exercises) for 50 minutes and local vibration applied to gastrocnemius (100 Hz) for 10 minutes will be performed 3 days a week for 8 weeks.
  Arms: Treatment Group 100 Hz
Other: Standard physiotherapy program — Standard physiotherapy program (strength, balance, gait exercises) for 60 minutes will be performed 3 days a week for 8 weeks.
  Arms: Control Group

SUMMARY:
Gastrocnemius spasticity is one of the main complaints in Multiple Sclerosis patients.Local muscle vibration is a method used for spasticity inhibition. However, when the studies in the literature are examined; It is noted that local vibration applications for spasticity are usually single sessions and evaluate the acute effect, do not produce functional outputs, there is no consensus on frequency and amplitude and the changes in muscle architecture are not examined. In this study, we aimed to investigate the effect of local vibration applied on spastic gastrocnemius on muscle architectural and functional properties in Multiple Sclerosis patients in addition to the standard physiotherapy program. The study was planned to include 3 groups, 2 treatment and 1 control group. The control group will receive standard physiotherapy, one of the treatment groups will receive 50 Hz local vibration in addition to standard physiotherapy, and other treatment group will receive 100 Hz local vibration in addition to standard physiotherapy. Disease severity, gastrocnemius spasticity, architectural and viscoelastic properties of muscle, ankle proprioception, balance and gait skills will be evaluated before and after 8 weeks treatment program. As a result; effectiveness of local vibration in addition to standard physiotherapy program and whether there is a difference between applications at different frequencies will be examined.

ELIGIBILITY:
Inclusion Criteria:

* > 18 years
* EDSS<5,5
* Gastrocnemius spasticity<2

Exclusion Criteria:

* having any injury or surgery of the lower extremity
* having systemic and metabolic disease
* having behavioral and cognitive problems that prevent consistence to guidelines given

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2019-12-15 (Actual); Primary Completion 2020-11 (Estimated); Study Completion 2020-12 (Estimated)

PRIMARY OUTCOMES:
Evaluation of Muscle Thickness and Fascicle Length with Ultrasonography | 3 minutes
  Bilateral Medial Gastrocnemius US evaluations were performed with use of a 5-10 MHz linear probe (Diasus Dynamic Imaging Ltd, Livingston, Scotland,UK). Patients were positioned prone position with their legs and their muscles relaxed for medial gastrocnemius. Muscle Thickness and Fascicle Length would be expressed as centimeters.
Evaluation of Pennation Angle with Ultrasonography | 2 minutes
  Bilateral Medial Gastrocnemius US evaluations were performed with use of a 5-10 MHz linear probe (Diasus Dynamic Imaging Ltd, Livingston, Scotland,UK). Patients were positioned prone position with their legs and their muscles relaxed for medial gastrocnemius. Pennation Angle would be angularly indicated.

SECONDARY OUTCOMES:
Assessment of spasticity | 5 minutes
  Modified Ashworth Scale (minimum score 0 (worse), maximum score 4 (better))
Assessment of viscoelastic properties of muscle | 5 minutes
  Myoton-3 (assessment of tone, elasticity and stiffness)
Assessment of ankle proprioception | 5 minutes
  Isokinetic dynamometer (Isomed 2000) (passive ankle joint position sense)
Assessment of single leg balance | 3 minutes
  Single leg balance test
Assessment of balance | 10 minutes
  Bertec Balance Check ScreenerTM force platform system (Assessment of limits of stability, anteroposterior and mediolateral sway range)
Assessment of gait characterictics | 5 minutes
  GAITRite Analysis System (assessment of velocity, step length, percentage of gait cycle spent in double and single support, stance phase, swing phase, base of support)

CONTACTS AND LOCATIONS:
Locations (1):
- Hacettepe University, Faculty of Physical Therapy and Rehabilitation, Ankara, Altındağ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ayvat F, Ozcakar L, Ayvat E, Aksu Yildirim S, Kilinc M. Effects of low vs. high frequency local vibration on mild-moderate muscle spasticity: Ultrasonographical and functional evaluation in patients with multiple sclerosis. Mult Scler Relat Disord. 2021 Jun;51:102930. doi: 10.1016/j.msard.2021.102930. Epub 2021 Mar 31. PMID 33836458